CLINICAL TRIAL: NCT06435767
Title: Quantitative Nodal Burden as a Determinant Identifying Ampullary Adenocarcinoma Patients Benefiting From Adjuvant Chemotherapy: A Retrospective Cohort Study
Brief Title: Quantitative Nodal Burden as a Determinant Identifying Ampullary Adenocarcinoma Patients Benefiting From Adjuvant Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dong Bing Zhao, Deputy director, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: CICAMS
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Ampullary Adenoma; Chemotherapy Effect
MeSH Terms: interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Adjuvant chemotherapy — In the Cancer Hospital, postoperative chemotherapy regimens and doses were planned by oncologists, with adjustments made based on drug toxicities or tumor responses.

SUMMARY:
Ampullary cancer, a rare malignancy, lacks standardized guidelines for effective multimodal treatment following curative resection. The opinions on whether postoperative chemotherapy can improve the long-term survival of ampullary adenocarcinoma (AA) are discordant. This aspect remains poorly studied, with comparably scant research conducted on it.

log odds of positive lymph nodes (LODDS), a quantitative variable, can continuously and accurately reflect the burden of nodal involvement, which suggested a potential ability to identify AA patients benefiting from postoperative adjuvant chemotherapy (ACT). Therefore, Mainly focused issues of ACT addressed in the study are as follows: 1) the role of ACT in improving long-term survival for patients with AA after curative resection. 2) the role of LODDS in identifying postoperative AA patients benefiting from ACT. 3) compared with T and N classifications reported previously, the advantage of LODDS in identifying ACT-benefited patients.

In this cohort study, a large scale of sample size was conducted by drawing on the collective experience of the National Cancer Center of China. The patients treated with radiotherapy were excluded to concentrate on the effect of ACT.

ELIGIBILITY:
Inclusion Criteria:

Pathologically confirmed AA patients without distant metastasis treated with curative-intent resection

Exclusion Criteria:

patients who received neoadjuvant therapy or radiotherapy, as well as those with missing clinical pathological or follow-up information

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In this international, retrospective cohort study, the cohort of Chinese enrolled patients who underwent curative surgery for AA at the National Cancer Center of China, Chinese Academy of Medical Sciences, Cancer Hospital, from January 1, 1998, to December 31, 2020 (NCC cohort). The Ethics Committee of the National Cancer Center of China approved the study. Informed consent was secured from participants, authorizing the utilization for potential research. Additionally, patients with AA between January 1, 2004, and December 31, 2017, in the surveillance, epidemiology and end results program were collected as the Western cohort. In which, 12 registries were enrolled including Alaska Natives, California, Connecticut, Georgia, Hawaii, Iowa, Kentucky, Louisiana, New Jersey, New Mexico, Seattle (Puget Sound), and Utah.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The role of adjuvant chemotherapy(ACT) | 1 year
  The association between ACT and Overall Survival (OS) of patients

SECONDARY OUTCOMES:
The role of adjuvant chemotherapy(ACT) | 1 year
  The association between ACT and Cancer-specific Survival (CSS) of patients
The role of adjuvant chemotherapy(ACT) | 1 year
  The association between ACT and Recurrence-free Survival (RFS) of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic and Gastric Surgical Oncology, National Cancer Center/ National Clinical Research for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China